CLINICAL TRIAL: NCT01070095
Title: The Electronic Asthma Action Plan System for Implementation in Primary Care
Acronym: eAAPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 10-052
Record Dates: First submitted 2010-02-16; First posted 2010-02-17 (Estimated); Results first posted 2019-09-13 (Actual); Last update posted 2019-09-13 (Actual); Status verified 2019-09

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Electronic Asthma Action Plan System (Experimental): Electronic Asthma Action Plan System (eAAPS)
  Interventions: Other: Electronic Asthma Action Plan System

INTERVENTIONS:
Other: Electronic Asthma Action Plan System — The electronic asthma action plan system consists of a tablet device in the physician waiting room which participants use to complete a simple questionnaire, a computerized clinical decision support system which then processes these data to produce a set of asthma care recommendations for the clinician, and finally, a printable asthma action plan that is given to patients, along with the URL for an asthma education website.

SUMMARY:
Asthma is a common and potentially fatal chronic disease. An asthma action plan (AAP) is a written plan produced by a physician for a patient with asthma, to provide education and guidelines for self-management of worsening asthma symptoms. Studies have shown that AAPs effectively improve asthma control, but physicians fail to provide AAPs due to lack of time and adequate skills. Physicians also often fail to determine if their patients have good asthma control, and to adjust medications in response to patients' control level. The investigators propose to develop and test a computerized tool that will help physicians to determine if their patients' asthma is well controlled, advise them on medication changes required according to the current level of control, and automatically generate an electronic version of the AAP, all based on patient responses to a questionnaire. The investigators hope that this system will eliminate the barriers that physicians face in determining asthma control, adjusting medications, and delivering an AAP, and will increase the frequency with which physicians are able to achieve these goals in patients with asthma. The objectives of the study are to determine the impact of this system on asthma action plan delivery by primary care physicians, the frequency of checking control level, and the frequency and appropriateness of asthma medication changes (in accordance with control). We will also attempt to determine the impact of the system on hospitalisations, emergency room (ER) visits, unscheduled visits to the doctor, total visits to the doctor, days off work or school, nocturnal asthma symptoms, daytime asthma symptoms, daytime rescue puffer use, and quality of life, and to measure physicians' perceptions of and satisfaction with the system.

DETAILED DESCRIPTION:
This is a 2-year prospective interrupted time series (ITS) study of usual asthma care (baseline period) (year 1) compared to care with the eAAPS in place (intervention period) (year 2). The setting is two academic family health teams (primary health care teams including family physicians, nurses, and allied health members) in Hamilton, Ontario and one community-based family health team in Brampton, Ontario.

ELIGIBILITY:
Inclusion Criteria:

* Eligible physicians will include all primary care physicians at the 4 sites.

Eligible patients will include:

* patients with asthma, as determined by a validated electronic chart record search algorithm for asthma and on an asthma medication [but not a Chronic Obstructive Pulmonary Disease (COPD) medication] within 1 year;
* patients >/= 16 years of age who understand English

Exclusion Criteria:

* Pregnant patients will be excluded given that conventional AAP recommendations may not be appropriate in this population.
* Any patient deemed to have cognitive limitations or a life expectancy of < 1 year

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2012-07; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samir Gupta, MDCM, Principal Investigator — Unity Health Toronto
Locations (3):
- Canada (3):
  - Wise Elephant Family Health Team, Brampton, Ontario
  - McMaster Family Health Team, Hamilton, Ontario
  - St. Michael's Hospital, Toronto, Ontario

REFERENCES:
- [Derived] Price C, Agarwal G, Chan D, Goel S, Kaplan AG, Boulet LP, Mamdani MM, Straus SE, Lebovic G, Gupta S. Large care gaps in primary care management of asthma: a longitudinal practice audit. BMJ Open. 2019 Jan 29;9(1):e022506. doi: 10.1136/bmjopen-2018-022506. PMID 30696669

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was carried out across two academic family health teams (primary health care teams including family physicians, nurses, and allied health members) in Hamilton, Ontario and one community-based family health team in Brampton, Ontario. Clinics used the OSCAR electronic medical record (EMR) system and were under a capitated funding model.
Pre-assignment Details: Only clinicians/practitioners were enrolled in the trial, but data were collected from patients of the clinicians so they are represented as a separate group. All asthma patients of enrolled clinicians were included in the analysis, but patients seen in the baseline/intervention periods were not necessarily the same and their number thus differs.
Groups:
- Electronic Asthma Action Plan System - Clinicians: All clinicians who consented to the study, who were invited to use the electronic asthma action plan system for their eligible patients
- Electronic Asthma Action Plan System - Patients: Eligible patients from clinicians who consented to the study
Period: Baseline Period
Arm/Group | Electronic Asthma Action Plan System - Clinicians | Electronic Asthma Action Plan System - Patients
Started | 19 | 830
Completed | 18 | 830
Not Completed | 1 | 0
Period: Intervention Period
Arm/Group | Electronic Asthma Action Plan System - Clinicians | Electronic Asthma Action Plan System - Patients
Started | 18 | 890
Completed | 18 | 890
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The total number of unique patients across the two periods entered; data on clinician demographics were not captured exclusively for the 18 consenting clinicians
Groups:
- Electronic Asthma Action Plan System - Patients: All eligible unique patients from clinicians who consented to the study
Arm/Group | Electronic Asthma Action Plan System - Patients
Number analyzed (Participants) | 1272
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: 830 eligible patients were seen in the baseline period and 890 seen in the intervention period. There were 1272 unique patients seen over the study period, with 382 (30.0%) seen exclusively in the baseline period, 442 (34.8%) seen exclusively in the intervention period, and 448 (35.2%) seen in both periods.
  years
    Baseline Period Age: number analyzed (Participants) | 830
    Baseline Period Age | 45.9 (17.4)
    Intervention Period Age: number analyzed (Participants) | 890
    Intervention Period Age | 47.3 (17.2)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 830 eligible patients were seen in the baseline period and 890 seen in the intervention period. There were 1272 unique patients seen over the study period, with 382 (30.0%) seen exclusively in the baseline period, 442 (34.8%) seen exclusively in the intervention period, and 448 (35.2%) seen in both periods.
  Participants
    Baseline Period Sex: number analyzed (Participants) | 830
    Baseline Period Sex: Female | 602
    Baseline Period Sex: Male | 228
    Intervention Period Sex: number analyzed (Participants) | 890
    Intervention Period Sex: Female | 632
    Intervention Period Sex: Male | 258

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants to Whom an AAP (Asthma Action Plan) Was Delivered by the Clinician
Description: Number of eligible patients to whom an AAP was delivered by the physician during the intervention period (52 weeks) compared to the baseline period (52 weeks) Predictor model to include: clinic, appointment provider practitioner type, prior objective diagnosis of asthma, documented physician diagnosis of asthma, presenting complaint type, billing physician (most responsible physician/other), previous emergency department (ED) visits/hospitalizations for asthma, and current asthma control
Time Frame: 24 months
Population: Number of patients on an asthma controller medication [either inhaled corticosteroid (ICS), ICS/long-acting beta agonist (LABA), or leukotriene receptor antagonist (LTRA)] for at least 1 visit in the study period, who received an AAP, and had not received/reviewed an asthma action plan in the last 6 months (a subset of the intervention population).
Measure: Count of Participants; unit: Participants
Groups:
- Baseline Period: 12 months pre-intervention
- Intervention Period: 12 months post-intervention (eAAPS)
Arm/Group | Baseline Period | Intervention Period
Number analyzed (Participants) | 412 | 443
Participants | 0 | 79

2. Secondary Outcome: The Impact of the eAAPS on Patient-relevant Outcomes Including Hospitalisations, Emergency Room Visits, Unscheduled & Total Visits to the Doctor, Days Off Work/School, Nocturnal/Daytime Asthma Symptoms, Daytime Rescue Bronchodilator Use & Quality of Life.
Time Frame: Every 2 weeks for 6 months
Population: Not measured due to inadequate patient outcome measurement recruitment
Arm/Group | Baseline Period | Intervention Period
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Asthma Control Assessment
Description: The number of patients with asthma control determined at least once, according to symptom-based criteria (control determination required meeting one or more criteria for uncontrolled asthma or all criteria for controlled asthma).
  Predictor model to include: clinic, appointment provider practitioner type, prior objective diagnosis of asthma, documented physician diagnosis of asthma, presenting complaint type, billing physician (most responsible physician/other), previous emergency department (ED) visits/hospitalizations for asthma, and current asthma control
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Baseline Period | Intervention Period
Number analyzed (Participants) | 830 | 890
Participants | 118 | 523

4. Secondary Outcome: Medication Escalations
Description: The number of patients with escalation of controller therapy Predictor model to include: clinic, appointment provider practitioner type, prior objective diagnosis of asthma, documented physician diagnosis of asthma, presenting complaint type, billing physician (most responsible physician/other), previous emergency department (ED) visits/hospitalizations for asthma, and current asthma control
Time Frame: 24 months
Population: In the measuring therapy escalation, we eliminated visits in which patients had had a controller medication escalated within the last three months (the typical duration of a therapeutic trial)
Measure: Number; unit: participants
Arm/Group | Baseline Period | Intervention Period
Number analyzed (Participants) | 830 | 890
participants | 106 | 117

5. Secondary Outcome: Appropriate Medication Changes
Description: Number of eligible visits in which patients who had an appropriate medication change made (i.e. escalation for poor control, and de-escalation for good control, when ascertainable)
Time Frame: 24 months
Measure: Number; unit: Visits
Units Other Than Participants: Visits
Arm/Group | Baseline Period | Intervention Period
Number analyzed (Participants) | 830 | 890
Number analyzed (Visits) | 3563 | 3327
Visits | 113 | 85

6. Secondary Outcome: On Treatment Analysis
Description: Number of eligible patients to whom an asthma action plan (AAP) was delivered, when decision support was available (52 weeks), counting only intervention period visits in which patients completed the questionnaire before the appointment and the notification prompted clinicians to open the computerized clinical decision support system (CDSS) to take action
Time Frame: During the 12 month intervention period
Population: Number of eligible patients with AAP delivery. This counts only patients for whom a prompt was presented to the clinician, so is a subset of the intervention population. We have only presented data from the Intervention Period, as this outcome pertains to the uptake of the intervention, and is not applicable to the Baseline Period.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Period
Number analyzed (Participants) | 265
Participants | 81

7. Secondary Outcome: Number of Practitioners Completing Feedback Questionnaires
Description: Number of practitioners completing feedback questionnaires on the system (delivered in the 1 month after end of intervention period)
Time Frame: 13 months
Population: Responding physicians. We have only presented data from the Intervention Period, as questionnaires were provided after the intervention only.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Period
Number analyzed (Participants) | 18
Participants | 12

8. Secondary Outcome: Ratio of Rescue to Controller Medication Prescriptions
Description: Ratio of rescue to controller medication prescriptions made during baseline vs intervention periods
Time Frame: 24 months
Measure: Number; unit: Ratio of SABAs to controllers prescribed
Arm/Group | Baseline Period | Intervention Period
Number analyzed (Participants) | 830 | 890
Ratio of SABAs to controllers prescribed | 1.15 | 0.14

9. Secondary Outcome: Adherence Discussions
Description: The number of patients in the intervention period in whom discussions about medication adherence took place
Time Frame: During the 12 month intervention period
Population: We have only presented data from the Intervention Period, as this was not captured in the Baseline Period.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Period
Number analyzed (Participants) | 890
Participants | 219

10. Secondary Outcome: System Uptake
Description: Actual usage of the system: number of patients for whom clinicians accessed the CDSS when actions were required
Time Frame: During the 12 month intervention period
Population: Number of patients for whom clinicians accessed the CDSS when actions were required based on the information entered in the questionnaire (a subset of the total intervention group). We have only presented data from the Intervention Period, as this outcome pertains to the uptake of the intervention, and is not applicable to the Baseline Period.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Period
Number analyzed (Participants) | 505
Participants | 174

ADVERSE EVENTS:
Description: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed in physicians or patients with asthma at any time point during the study. This was a quality improvement study, with a tool to improve clinician practice. As such, participants were not considered at risk.
Groups:
- Baseline: 12 months pre-intervention
- Intervention: 12 months post-intervention (eAAPS)
Arm/Group | Baseline | Intervention
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
An interrupted time series design is vulnerable to temporal factors that may have affected asthma care behaviour. We report on behavioural rather than health outcomes in this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No